CLINICAL TRIAL: NCT02729012
Title: Effects of Hypertonic Saline Solution (NACL 3%+NAHCO3) on Nasal Inflammation in Children With Allergic Rhinitis. RinASol- Pilot Study (Allergic Rhinitis Solution)
Brief Title: Effects of Hypertonic Saline Solution (NACL 3%+NAHCO3) on Nasal Inflammation in Children With AR. RinASol- Pilot Study
Acronym: RinASol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: -11/2014
Record Dates: First submitted 2016-03-04; First posted 2016-04-06 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Allergic Rhinitis
Keywords: Children
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Saline Solution, Hypertonic; Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case (Active Comparator): Allergic Rhinitis Children treated with hypertonic saline solution (NACL 3%+NAHCO3)
  Interventions: Drug: hypertonic saline solution (NACL 3%+NAHCO3)
- Control (Placebo Comparator): Allergic Rhinitis Children treated with saline solution (NACL 0,9%)
  Interventions: Other: Saline Solution (NACL 0,9%)

INTERVENTIONS:
Drug: hypertonic saline solution (NACL 3%+NAHCO3) — Treatment with nebulized hypertonic saline solution (NACL 3%+NAHCO3)
  Arms: Case
Other: Saline Solution (NACL 0,9%) — Treatment with nebulized Saline Solution (NACL 0,9%)
  Arms: Control

SUMMARY:
The main objective of RinASol project is to assess in patients with seasonal Allergic Rhinitis the effect of hypertonic saline solution NACL 3%+NAHCO3 vs the effect of standard saline solution on nasal inflammation by means of nasal cytology.

The secondary objective is the symptom score assessment by T5SS Questionnaire (Total Symptom Score 5)

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of Allergic Rhinitis (for at least 1 year)
* 6 years old ≤ children age ≤ 14 years old
* Total Symptom Score 5: >5 in the last 4 days before screening. Exclusion Criteria
* Signs of acute infections of upper and lower respiratory tract.
* Metabolic, immunological, systemic diseases
* Respiratory tract deformity
* Systemic/Topical therapies with antibiotics or corticosteroids in the previous 30 days.
* Active smoker.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Symptom score assessment | 28 days
  The main objective is to evaluate the effect of hypertonic saline solution NACL 3%+NAHCO3 vs the effect of standard saline solution on the symptom score assessed by T5SS Questionnaire (Total Symptom Score 5)

SECONDARY OUTCOMES:
Nasal cytology pattern | 28 days
  The secondary objective is to evaluate the effect of hypertonic saline solution NACL 3%+NAHCO3 vs the effect of standard saline solution on nasal inflammation, in patients with seasonal Allergic Rhinitis, by means of nasal cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania La Grutta, MD, Principal Investigator — IBIM,CNR, PALERMO, ITALY
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No